CLINICAL TRIAL: NCT06781437
Title: Studio Osservazionale Retrospettivo Di Coorte Italiana Di Pazienti Con Linfoma (RETRO-LYMPH)
Brief Title: Retrospective Observational Study of Italian Cohort of Lymphoma Patients (RETRO-LYMPH)
Acronym: RETRO-LYMPH
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: RETRO-LYMPH
Record Dates: First submitted 2024-12-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Lymphoproliferative Syndrome, Autoimmune; Lymphoma
MeSH Terms: conditions — Autoimmune Lymphoproliferative Syndrome; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
observational, non-interventional, retrospective, single-center study focusing on patients with lymphoma / lymphoproliferative syndrome between January 1980 and September 2021

DETAILED DESCRIPTION:
observational, non-interventional, retrospective, single-center study focusing on patients with lymphoma / lymphoproliferative syndrome between January 1980 and September 2021.

Study objectives are to enrich the data on the prognostic role of clinical and epidemiological factors associated with clinical and epidemiological data of patients;

* to identify the factors that affect the evolution of the disease, such as lifestyle and occupational factors, as well as the type of treatment;
* to provide a platform for future research projects;
* Description of the various therapies that have occurred over time, duration of treatment, causes of interruption of treatment, responses;
* Description of the adverse events / safety of the various therapies for lymphoma and lymphoproliferative syndromes;
* Patient survival. Descriptive analyses will be conducted by tabulating frequency distributions and percentages and mean and median values, standard deviations, quartiles and extreme values for continuous variables. Progression-free survival, disease-free survival and overall survival will be examined using Kaplan-Meier point estimates

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of enrollment
* Diagnosis of lymphoma or lymphoproliferative syndrome between January 1980 and September 2021
* Signature of the informed consent form where applicable

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lymphoma / lymphoproliferative syndrome between January 1980 and September 2021
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and prevalence of lymphomas/lymphoproliferative syndromes referred to the Centre between January 1980 and September 2021 | through study completion, an average of 6 years
  Incidence and prevalence

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 6 years
  Overall Survival (OS)
event free survival (EFS) | through study completion, an average of 6 years
  event free survival (EFS)
Lymphoma specific survival (LSS) | through study completion, an average of 6 years
  Lymphoma specific survival (LSS)
Progression Free Survival (PFS) | through study completion, an average of 6 years
  Progression Free Survival (PFS)
Net survival (5 years) | through study completion, an average of 6 years
  Net survival
Response rate (5 years) | through study completion, an average of 6 years
  Response rate
Duration of Response (DoR) | through study completion, an average of 6 years
  Duration of Response (DoR)
time to next anti-lymphoma treatment (TTNLT) | through study completion, an average of 6 years
  time to next anti-lymphoma treatment (TTNLT)
Duration of survival after progression | through study completion, an average of 6 years
  Duration of survival after progression
lymphoma transformation frequency | through study completion, an average of 6 years
  lymphoma transformation frequency
Frequency of secondary neoplasy | through study completion, an average of 6 years
  Frequency of secondary neoplasy
frequency of other chronic diseases | through study completion, an average of 6 years
  frequency of other chronic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No